CLINICAL TRIAL: NCT05131503
Title: Evaluation of The Fear of Childbirth in Pregnant Women Who Are In The Antenatal Polyclinic: The Sample of Turkey
Brief Title: Evaluation of The Fear of Childbirth
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nükhet Kaçar, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkent-MH-NK-02
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Fear of Childbirth
Keywords: fear; Parturition; midwifery; Pregnant Women

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Research — Non-applicable. There is no intervention. This study is descriptive research.

SUMMARY:
Most pregnant women have fear of labor. The reasons of fear of labor are different according to women. The investigators will examine the relationship between the descriptive features and level of fear of labor of pregnant women by using the Oxford worries about labour scale

DETAILED DESCRIPTION:
The investigators will give a survey to pregnant women who go to the antenatal polyclinic. The survey is consisted by researchers. The survey has a few questions about pregnant women's descriptive features. Next the investigators will evaluate the level of fear of labor of pregnant women. After the investigators will analyze the relationship between pregnant women's fear and their descriptive features.

ELIGIBILITY:
Inclusion Criteria:

* all of volunteers and pregnant women who are 18-35 years old.

Exclusion Criteria:

* the pregnant women have any obstetrical complications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We will study with pregnant women.
Study Population: they are healthy pregnant women who are 18-35 years old. they do not have any obstetrical complications. they go to the antenatal polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
The Oxford Worries About Labour Scale | approximately 30 minutes, waiting in the antenatal polyclinic.
  This scale measures the level of fear of childbirth. The scale has ten questions which has four answers as Likert Scale. Also the scale has 40-100 points. As the point decreases the fear score increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nükhet Kaçar, MSc., Principal Investigator — Ankara City Hospital- Maternity Hospital
Locations (1):
- Ankara City Hospital- Maternity Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No